CLINICAL TRIAL: NCT01627496
Title: Nutritional Status and Quality of Life in Older Hospitalised Adults
Brief Title: Nutritional Status and Quality of Life in Older Adults
Acronym: NSQLOP
Status: Completed | Type: Observational
Sponsor: University of Surrey (Other)
Responsible Party: Principal Investigator, Kathryn Hart, Lecturer in Nutrition & Dietetics, University of Surrey
Other Study IDs: NSQLOP
Record Dates: First submitted 2012-06-15; First posted 2012-06-25 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Malnutrition
Keywords: malnutrition; elderly care; quality of life; hospital
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to determine the nutritional status, and factors affecting malnutrition in older people staying in hospitals.

Objectives:

* To recruit a sample of older people in hospital
* To collect information on nutritional status, satisfaction with food-related life and experience with access to food in hospital.
* To assess the staffing attitudes to nutritional care of the older adult
* To undertake an audit of therapeutic ('special') diets served in hospitals, with respect to their nutritional adequacy and wastage
* To investigate predictors and correlates of malnutrition within the hospital setting and compare these relationships with those previously identified in care homes and the community.
* To make recommendations for practice to improve the nutritional status of hospitalised older adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 75 years old
* Male or female
* Duration of stay is more than 24hrs
* Able to eat normally
* Able to read and write English
* Able to be weighed standing or sitting OR accurate weight available since admission

Exclusion Criteria:

* Age below 75 years old
* Newly admitted patient (less than 24hrs)
* Certain medical conditions likely to affect digestion/ absorption of nutrients (researchers will assess)
* Unable to provide informed written consent
* Patients on gastric surgical wards or suffering from gastritis
* Patients currently taking laxatives
* Unable to be weighed and no measured weight available (self report weight is not adequate)

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Hospitalised older adults (>75years)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Nutritional status | baseline
  Using MNA
Satisfaction with food related quality of life | baseline
Dietary intake | baseline
  3 x 24hr recalls

SECONDARY OUTCOMES:
Food Access in Hospital | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Noraida Omar, BSc, Principal Investigator — University of Surrey
Locations (1):
- Royal Surrey County Hospital, Guildford, Surrey, United Kingdom